CLINICAL TRIAL: NCT00901264
Title: Correlation of the Microculture Kinetic (MiCK) Apoptosis Test Results With Drug Treatment Results in Cancer Patients
Brief Title: Microculture Kinetic (MiCK) Apoptosis Test Results With Drug Treatment Results in Cancer Patients
Acronym: MiCK
Status: Completed | Type: Observational
Sponsor: Pierian Biosciences (Industry)
Responsible Party: Sponsor
Other Study IDs: Master Study DiaTech Oncology
Record Dates: First submitted 2009-05-12; First posted 2009-05-13 (Estimated); Last update posted 2012-11-14 (Estimated); Status verified 2012-11

CONDITIONS: Cancer
Keywords: Chemosensitivity, chemotherapy, all cancers, personalized chemotherapy, personalized cancer treatment; Cancer Patients for whom chemotherapy is planned.
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- 1: Patients with pathological diagnoses of cancer or leukemia
- 2: 3.1.3 Patients for whom chemotherapy is planned.

SUMMARY:
The purpose of this study is to correlate the results of the MICK assay with short- and long-term results of treatments in cancer patients and evaluate the role of the MiCK assay in guiding chemotherapy of cancer patients.

DETAILED DESCRIPTION:
Identification of those patients with cancer who will or will not respond to a specific chemotherapy is important for making decisions regarding chemotherapy regimens as well as alternative management approaches. A laboratory test that could help to determine the sensitivity of an individual patient's tumor cells to specific chemotherapeutic agents would be valuable in choosing the optimal chemotherapy regimen for that patient with an expectation of increasing the response rate to the therapy. Several types of in vitro assays that measure tumor cell survival following exposure to cytotoxic agents have been evaluated for their ability to predict chemotherapy outcomes. As a group, these assays are referred to as drug resistance assays. In a resistance assay, the surviving tumor cells can be detected directly by their exclusion or metabolism of specific dyes. Alternatively, since some of tumor cells are proliferating, their survival can be detected by measurement of DNA synthesis by radiolabeled precursor incorporation or demonstration of clonogenic potential by growth into colonies in semi-solid culture medium. In several clinical studies, these assays were useful in detecting drug resistance and in predicting a poor prognosis for cancer patients. However, these resistance assays cannot detect sensitivity of an individual patient's tumor cells to a specific drug. Therefore, new methods determining drug-sensitivity of the tumor cells of an individual patient and, thus, capable of both predicting a positive treatment outcome and guiding chemotherapy, would be of significant value.

Recently, an automated microculture kinetic (MiCK) assay for measuring drug induced apoptosis in tumor cells has been developed1-4. Apoptosis is a distinct mode of cell death which occurs under physiological conditions and yet can be induced in malignant cells by chemical and physical factors including antitumor drugs5-7. During the last decade, it has been recognized that chemotherapeutic agents exert their antitumor activity by triggering apoptosis in susceptible tumor cells8-17. This implies that the MiCK assay for apoptosis provides a mechanism-based approach to studying effects of cytotoxic agents on tumor cells. Unlike "resistance" assays that measure a fraction of cells surviving drug exposure, the MiCK assay measures a fraction of tumor cells killed by a chemotherapeutic agent via mechanism of apoptosis. Therefore the MiCK assay determines drug sensitivity, rather than resistance. Recently the MiCK assay has been shown to predict complete remission rate and survival in acute myeloid leukemia patients better than clinical criteria did18-20. In a limited study, the MiCK assay has been used to direct chemotherapy of the leukemia patients 21.

The MiCK assay has also been used to study drug-induced apoptosis in solid tumors, including neuroblastoma and colon adenocarcinoma cell lines22-23. More recent data accumulated by DiaTech has demonstrated that the MiCK assay can detect drug induced apoptosis in primary cultures of tumor cells isolated from patients with ovarian carcinoma, gastric carcinoma, metastatic breast cancer and high grade soft tissue sarcoma. The purpose of this study is to correlate the results of the MICK assay with short- and long-term results of treatments in cancer patients and evaluate the role of the MiCK assay in guiding chemotherapy of cancer patients.

ELIGIBILITY:
Inclusion Criteria:

* 3.1.1 Patients with pathological diagnoses of cancer or leukemia
* 3.1.2 Patients must have tumor which is accessible for biopsy and agree to undergo tumor biopsy, or drainage of malignant effusion, and the specimen must be submitted for MiCK assay.
* 3.1.3 Patients for whom chemotherapy is planned.

Exclusion Criteria:

* 3.2.1 Patients with symptomatic/uncontrolled parenchymal brain or meningeal metastasis and tumors not accessible for biopsy.
* 3.2.2 Patients who are pregnant. Pregnancy. During the course of the study, all patients of childbearing potential should be instructed to contact the treating physician if they suspect they might have conceived a child; for females, a missing or late menstrual period should be reported to the treating physician. If pregnancy is confirmed by a pregnancy test, the patient must not receive chemotherapy in this study and must not be enrolled into the study or, if already enrolled, must be withdrawn from the study. If a male patient is suspected of having fathered a child while on the study, the pregnant female partner must be notified and counseled regarding the risk to the fetus. Pregnancy during the course of this study will be reported to the Principal Investigator as a serious adverse event. Women of child bearing potential are defined to include any female who has experienced menarche and has not undergone successful surgical sterilization (hysterectomy, bilateral tubal ligation, or bilateral oophorectomy) or is not post-menopausal (defined as amenorrhea for more than 12 consecutive months); these includes also females using oral, implanted, or injectable contraceptive hormones, mechanical devices, or barrier methods to prevent pregnancy.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Cancer Patients for whom chemotherapy is planned.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2008-12; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
To evaluate the ability of the MiCK assay to guide chemotherapy of cancer patients, with emphasis on patients failing primary treatment, patients with unknown primary tumors, and patients with tumors difficult to treat such as carcinoma of lung. | one year

SECONDARY OUTCOMES:
Correlate the MiCK assay results with objective response rates, symptom response rates, time to progression and survival of cancer patients treated with chemotherapy. | one year

CONTACTS AND LOCATIONS:
Overall Officials: Cary Presant, MD, Study Director — Pierian Biosciences; Dirk Davidson, MD, Principal Investigator — Cumberland Medical Center; Karl Rogers, MD, Principal Investigator — Nashville Oncology Associates; Swapnil P. Rajurkar, MD, Principal Investigator — Wilshire Oncology Medical Group, Inc.; Laura Lawson, MD, Principal Investigator — Tennessee Breast Specialists; L. James Wudel Jr., MD, Principal Investigator — Tennessee Thoracic Surgical Specialists; Raymond F Bluth, MD, Principal Investigator — Baptist Hospital Nashville; Peter F Jelsma, MD, Principal Investigator — St. Thomas Research Institute, LLC; Richard D Michaelson, MD, Principal Investigator — Middle Tennessee Medical Center; Jorge E Marcet, MD, Principal Investigator — Tampa Gerneral Hospital
Locations (11):
- United States (10):
  - Wilshire Oncology Medical Group, Inc, La Verne, California
  - Tampa General Hospital, Tampa, Florida
  - DiaTech Oncology, Brentwood, Tennessee
  - Cumberland Medical Center, Crossville, Tennessee
  - Middle Tennessee Medical Center, Murfreesboro, Tennessee
  - Baptist Hospital, Nashville, Tennessee
  - Nashville Oncology Associates, Nashville, Tennessee
  - St. Thomas Research Institute, LLC, Nashville, Tennessee
  - Tennessee Breast Specialists, Nashville, Tennessee
  - Tennessee Toracic Surgical Specialists, Nashville, Tennessee
- DiaTech Oncology, Montreal, Quebec, Canada

REFERENCES:
- [Derived] Bosserman L, Rogers K, Willis C, Davidson D, Whitworth P, Karimi M, Upadhyaya G, Rutledge J, Hallquist A, Perree M, Presant CA. Application of a drug-induced apoptosis assay to identify treatment strategies in recurrent or metastatic breast cancer. PLoS One. 2015 May 29;10(5):e0122609. doi: 10.1371/journal.pone.0122609. eCollection 2015. PMID 26024531